CLINICAL TRIAL: NCT06206213
Title: Investigation of the Effects of Two Types of Locomotion in the Virtual Environment in Terms of Postural Stability and Cybersickness.
Brief Title: Investigation of the Effects of Two Types of Locomotion in the Virtual Environment
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Çiğdem Yazıcı Mutlu, assistant prof, Yeditepe University
Other Study IDs: HMDs effect on body posture
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Cybersickness
Keywords: Postural Control; Virtual Reality; Locomotion

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy Young University Students: This study involves just one group which will be consist of 40 healthy young adults (university students). It will include both males and females and all of them will be exposed to the same protocol.
  Interventions: Behavioral: Assessment of two different locomotion types.

INTERVENTIONS:
Behavioral: Assessment of two different locomotion types. — Exposure to virtual environment by the HMD in two different locomotion styles.

SUMMARY:
Virtual Reality (VR) is a technology that enables individuals to engage in a computer-generated, three-dimensional (3D) environment by utilizing specialized electronic equipment. This technology allows users to explore and interact with a wide range of objects and events, enabling them to perform perspective and motor tasks (Frederick P. Brooks, 1999). VR head-mounted displays (HMDs) create full immersion in the virtual environment by projecting images on screens positioned very close to the eyes (Turnbull & Phillips, 2017).

The quick development of this technology has made it more affordable and available, consequently, its utilization is also increasing. It has applications in various fields, for example, it is widely used as a training platform for astronauts, soldiers, and treatment purposes in rehabilitation (Xie et al., 2021). The reason why many sectors urge to take advantage of VR is because they could promote motor learning by generating an environment, scenario, or activity that allows for the user practice motor skills with simple tools. Simultaneously, VR provides the possibility of repeating the same task at any moment, modifying factors such as level of complexity, time, and intensity of the practice (Lledó et al., 2016).

Despite the great expansion of virtual technology, cybersickness continues to be a problem that prevents it from being used fluently (Tian et al., 2022). Cybersickness is a term established to describe the unpleasant sensation that evokes from the use of virtual reality technology (McCauley & Sharkey, 1992). Cybersickness appears with symptoms like motion sickness symptoms, the ones we feel while using vehicle such as nausea, dizziness, fatigue, and blurred vision (Laviola, 2000). In various research studies, this phenomenon has been mentioned in different terms, such as simulator sickness or VR sickness. There are several theories trying to explain why individuals develop these symptoms when they are in the car or using HMDs, however, just two theories are considered the most accepted. First theory is the Sensory Conflict Theory that was proposed by Reason & Brand (1975) while the other one is the Postural Instability Theory, developed by Riccio & Stoffregen (1991).

There are several factors that affect the severity of cybersickness while using HMDs and some studies have already discussed them (Tian et al., 2022). One of the main factors in Interaction; Navigation method and controllability. Different locomotion styles, such as steering walking, or teleportation, have been investigated to the virtual environment for the purpose of navigating and showed that the choice of the locomotion style would heavily impact the user experience (Al Zayer et al., 2020).

From this point, our study is aiming to compare the difference between the most used locomotion style: controller-based steering, and the Walk in place (WIP), in the context of postural control and cybersickness. We are also planning to investigate other factors affecting the results, such as personal factors; gender, previous experience, and individual's susceptibility to motion sickness.

This study including healthy young volunteers (18-30-year-olds). They started to be collected from November 2023 and will continue until February 2024 in Yeditepe University Physiotherapy and Rehabilitation department laboratory.

Participants will be asked to fill in an online form or conduct a brief interview to collect their demographic information. They will be asked about their age, height (cm), weight (kg), body mass index (BMI), gender (female / male), Medical History, gaming experience, hand and leg preference and Susceptibility to motion sickness. Then, postural stability, motion sickness measurements and heart rate (HR) will be taken before and after each experimental trial.

All Participants will play a game called "Freedom locomotion VR" a 3D virtual environment allowing the player to do several activities in it. All participants will be immerged in this virtual environment twice (two sessions) and have the freedom to do what they like in it. However, In each session, they will use one the two locomotion types that the game provides, the hand controller (HC) based and walking in place (WIP) based locomotion. To compare the effect of each of the two locomotion styles, each participant will play the game two times to be able to try both locomotion types. Postural control, motion sickness symptoms and heart rate will be tested after each session to measure the different in the effect of each type of locomotion.

As this research is including one group who will be measured multiple times in the experiment, repeated measures one-way analysis of variance (ANOVA) would be the best statistical test to use to investigate the difference.

ELIGIBILITY:
Inclusion Criteria:

* Young Adults between 18 and 30 years old.
* Able to understand and follow the researchers' instructions.
* Have no pain or any medical illness.
* Have normal or corrected to normal vision.
* Volunteering to participate in experiments.

Exclusion Criteria:

* Having any medical problem that could affect physical movement or balance (e.g., vestibular, sensory, or musculoskeletal impairments)
* Having any visual problems.
* Having any neurological disorder.
* Using an additional assistive device.
* Have had a middle ear infection in the past month.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy university students who are aged between 18 to 30.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Assessment of Simulator Sickness symptoms: Simulator Sickness Questionnaire (SSQ) | 2 minutes
  Simulator Sickness Questionnaire (SSQ) is a short questionnaire that use to evaluate the symptoms occur with the exposure of virtual reality. It is used to determine the severity of simulator sickness symptoms by giving a score of 16 different items. The severity of each symptom in this questionnaire is measured on a four-point scale (0 = Not at all, 1 = Mild, 2 = Moderate, 3 = Severe). Symptoms in SSQ are determined according to the severity of 3 main factors:
  Nausea (such as sweating, difficulty concentrating, stomach awareness) Oculomotor Disturbances (such as headache, eyestrain, blurred vision) Disorientation (head fullness, eyesight, dizziness, vertigo)
Assessment of Postural Control: Prokin PK 252, the proprioceptive-stabilometric assessment device | 10 min
  The Prokin device (Prokin PK 252) is a proprioceptive system used for static and dynamic balance assessment and training. For this experiment, "Static Stability Assessment Program" will be chosen to provide detailed and precise data of each participant while static standing through the stabilometry platform. Stabilometry allows participants to be evaluated by detecting the oscillation of the Centre of Pressure (CoP) during static standing.

SECONDARY OUTCOMES:
Assessment of Motion sickness susceptibility: The motion sickness susceptibility questionnaire - Short form (MSSQ-Short) | 2-3 minutes
  MSSQ is used to evaluate the participants' susceptibility to motion sickness. The questionnaire asks about signs of feeling uncomfortable, nausea, and vomiting in different situations to determine which type of movement is causing motion sickness. The participants will answer according to their previous experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem Yazici Mutlu, PhD, Study Director — Yeditepe University
Locations (1):
- Yeditepe university, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brooks FP. What's real about virtual reality?. IEEE Computer graphics and applications. 1999 Nov;19(6):16-27.
- [Background] Turnbull PRK, Phillips JR. Ocular effects of virtual reality headset wear in young adults. Sci Rep. 2017 Nov 23;7(1):16172. doi: 10.1038/s41598-017-16320-6. PMID 29170432
- [Background] Xie B, Liu H, Alghofaili R, Zhang Y, Jiang Y, Lobo FD, Li C, Li W, Huang H, Akdere M, Mousas C. A review on virtual reality skill training applications. Frontiers in Virtual Reality. 2021 Apr 30;2:645153.
- [Background] Lledo LD, Diez JA, Bertomeu-Motos A, Ezquerro S, Badesa FJ, Sabater-Navarro JM, Garcia-Aracil N. A Comparative Analysis of 2D and 3D Tasks for Virtual Reality Therapies Based on Robotic-Assisted Neurorehabilitation for Post-stroke Patients. Front Aging Neurosci. 2016 Aug 26;8:205. doi: 10.3389/fnagi.2016.00205. eCollection 2016. PMID 27616992
- [Background] Tian N, Lopes P, Boulic R. A review of cybersickness in head-mounted displays: raising attention to individual susceptibility. Virtual Reality. 2022 Dec;26(4):1409-41.
- [Background] McCauley ME, Sharkey TJ. Cybersickness: Perception of self-motion in virtual environments. Presence: Teleoperators & Virtual Environments. 1992 Aug 1;1(3):311-8.
- [Background] LaViola Jr JJ. A discussion of cybersickness in virtual environments. ACM Sigchi Bulletin. 2000 Jan 1;32(1):47-56.
- [Background] Reason, J.T. and Brand, J.J., 1975. Motion sickness. Academic press.
- [Background] Riccio GE, Stoffregen TA. An ecological theory of motion sickness and postural instability. Urbana. 1991;100:6180.
- [Background] Al Zayer M, MacNeilage P, Folmer E. Virtual Locomotion: A Survey. IEEE Trans Vis Comput Graph. 2020 Jun;26(6):2315-2334. doi: 10.1109/TVCG.2018.2887379. Epub 2018 Dec 18. PMID 30575541